CLINICAL TRIAL: NCT02673957
Title: Analysis of Local and Circulating Compounds Released Following Hypoxia Induced by Blood Pressure Cuff Inflation
Brief Title: Analysis of Local and Circulating Compounds Released Following Blood Pressure Cuff Inflation
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn
Sponsor: University of New England, Australia (Other)
Responsible Party: Principal Investigator, Jacqueline Epps, Dr Jacqueline Epps, University of New England
Other Study IDs: HE15-280
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral venous blood samples, which are processed by centrifuge. The plasma will be extracted and retained for analysis, with the rest of the sample discarded.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood pressure cuff protocol: All participants receive a baseline control blood test, and all participants receive the blood pressure cuff inflation protocol and blood sampling following the cuff protocol.
  Interventions: Other: Blood pressure cuff protocol

INTERVENTIONS:
Other: Blood pressure cuff protocol — 4 cycles of pneumatic blood pressure cuff inflation to 200mmHg for 5 minutes followed by 5 minutes of deflation. Each subsequent cycles commences as soon as the previous cycle is completed.

SUMMARY:
This study aims to analyze the way the human body responds to a temporary lack of oxygen, or ischaemia. Prospective participants will complete a health screen to confirm overall health / low cardiovascular risk profile.The participants will be required to have pneumatic blood pressure cuff inflation to 200mmHg on the upper arm for 5 minutes which will then be deflated for 5 minutes and then repeating the cycle of inflation and deflation a further 3 times. Blood tests from veins in the forearm would be taken before, during, and after this is done in order to compare results and establish any change in concentration of local and circulating compounds.

DETAILED DESCRIPTION:
Evidence exists that short periods of ischaemia (lack of oxygen delivered to tissue in the body) can protect a local or remote area of the body from subsequent prolonged periods of serious ischaemia. It has been shown that substances are released into the circulation after short periods of ischaemia that may cause this protection. This study aims to identify some of these compounds.

After participants are informed about the study and have an opportunity to ask questions, informed consent will be obtained. Following this, a modified Exercise and Sports Science Australia questionnaire and brief medical history will be obtained. Blood pressure readings, height, weight and waist circumference would be measured. This is to establish a picture of overall general health and cardiovascular risk profile.

Those who meet the study eligibility criteria will proceed on a subsequent day to the blood pressure cuff inflation protocol. Consumption of caffeine or alcohol cannot be consumed within 4 hours prior to the protocol and participants must minimise any physical activity in the 4 hours prior to the protocol. After resting for 15 minutes on arrival, a baseline venous blood test will be taken from the dominant arm. A standard pneumatic blood pressure cuff will be placed around the non-dominant upper arm and inflated to 200mmHg for 5 minutes. The cuff will then be deflated completely for 5 minutes. This cycle will be repeated a further 3 times, with each cycle commencing as soon as the previous one has been completed. At the end of the final deflation, a second venous blood sample will be taken from the arm with the cuff. 10 minutes after this, a final venous blood test will be taken from the dominant arm. Blood samples will be processed and stored appropriately until analysed by mass spectrometry. Changes in compounds in the cuffed limb and the opposite limb from the baseline blood sample will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* healthy with no known chronic medical conditions
* low cardiovascular risk
* no recent significant illness or injury
* able to provide informed consent

Exclusion Criteria:

* pregnancy or breastfeeding
* moderate or high cardiovascular risk
* chronic medical condition
* taking regular or recent medication, including herbal remedies, recreational drugs or over-the-counter medication
* smoking within the previous 12 months
* previous or current vascular disorders including deep vein thrombosis
* bleeding disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes in local and circulating compounds following blood pressure cuff occlusion protocol | Last blood sample collected 10 minutes following completion of protocol
  Extracted plasma from venous blood samples will be analyzed by mass spectrometry to assess for any changes when compared with baseline blood test

CONTACTS AND LOCATIONS:
Overall Officials: Neil Smart, PhD M.Med Sci, Study Chair — University of New England
Locations (1):
- University of New England, Armidale, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No